CLINICAL TRIAL: NCT03989999
Title: Transcranial Ultrasonography for the Management of Patients With Mild Traumatic Brain Injury
Brief Title: Transcranial Ultrasonography for the Management of Patients With Mild TBI
Acronym: TRUST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 38RC19.106
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Transcranial Doppler
MeSH Terms: conditions — Brain Concussion | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open, non-inferiority, randomized, controlled, study with blinded evaluation.
Who Masked: Outcomes Assessor
Masking Description: The evaluation at 3 months after TBI will be centralized by the coordinating centre and blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TCD Group (Experimental): Transcranial Doppler within 12 hours of traumatic injury
  Interventions: Procedure: Transcranial Doppler (TCD)
- CONTROL Group (No Intervention): Mild TBI management with SFMU recommandations

INTERVENTIONS:
Procedure: Transcranial Doppler (TCD) — In the Emergency Department (ED):
  After the initial cerebral CT scan, the patient will be included in the study when he/she satisfies inclusion criteria. TCD will be performed within 12 hours of the brain injury.
  If TCD is normal (FVd>25 cm/sec and PI <1.25), the patient will return home under third-party supervision. An advice sheet will be given to the patient according to the SFMU guidelines and another one will be sent to the general practitioner. If initial cerebral CT scan is performed early (< 4-6 hours after TBI), CT scan should not be controlled before patient discharge.
  If the TCD is abnormal (FVd≤25 cm/sec or PI ≥ 1.25) the patient will be hospitalized. There is no recommendation regarding the type of hospitalization (ICU or standard ward).
  No other diagnostic procedure is allowed in the ED (S-100 protein dosing is not allowed). All therapies recommended by the SFMU for mild TBI are allowed in this group.
  Arms: TCD Group

SUMMARY:
The investigators hypothesize that patients with mild TBI and normal TCD can be safely discharged home immediately after the ED. The targeted population is the category of patients eligible for early discharge: 1) patients with mild lesions on the initial CT scan and a GCS 15 after CT scan completion and, 2) patients with no lesion on the initial cerebral CT scan with at least one of the following risk factors: GCS 14 after CT scan completion, persisting post-traumatic nausea/vomiting/headaches, concomitant alcoholic intoxication or patients treated with aspirin. The study will not include mild TBI patients who are not eligible for early discharge: patients with no possibility of home supervision, those with a GCS lower than 14 after the CT scan or those treated with anticoagulant/antiplatelet drugs other than aspirin. The investigators expect the TCD-based strategy to be non-inferior compared to the standard strategy according to French recommendations in terms of the 3-months neurological outcome. From a public health standpoint, the use of TCD as a triage tool may change current guidelines regarding mild TBI management.

DETAILED DESCRIPTION:
Patients with mild traumatic brain injury (TBI) represent the vast majority of TBI patients admitted in the emergency department (ED). According to French recommendations, mild TBI patients with brain lesions on initial CT scan are directed to a standard ward, where neurologic monitoring consists of repeated CT scanning and clinical exams. Patients with no lesion on initial cerebral CT scan are also hospitalized 1) when their GCS after CT scan is lower than 15, 2) in case of persisting nausea, vomiting or headache, 3) in case of concomitant alcoholic intoxication and, 4) in case of on-going treatment with aspirin. This strategy induces significant hospital stay with potential morbidity, whereas neurologic worsening rarely occurs.

In this context, the implementation of a triage tool in the ED would be useful to screen patients at risk of early neurologic worsening. Hence, low risk patients may be discharged at home immediately after the ED. Transcranial Doppler (TCD) is a non-invasive technique that measures cerebral blood flow velocities in intracranial cerebral arteries. These velocities and a derivated parameter (pulsatility index, PI), estimate cerebral blood flow (CBF) and have become a standard of care to optimize CBF in after severe TBI. Only few studies report the use of TCD after mild TBI. In a single-center cohort of patients with mild-to-moderate TBI, TCD parameters measured at hospital admission accurately predicted early neurologic worsening. These encouraging results indicate that TCD, in combination with CT scan findings, could play a role in the management of patients with mild TBI.

The aim of this project is to determine whether a TCD-based strategy is non-inferior to the standard management in terms of the overall neurological outcome at 3 months after mild TBI with no/minor lesions detected on a cerebral CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Mild TBI (GCS 13-15 on ED admission) with one of the following:
* Patient with minor cerebral lesion on initial CT scan (TCDBII i.e. no midline shift, visible basal cisterns and haemorrhagic lesion < 25 cc) and GCS 15 after CT scan
* OR * Patient with normal initial CT scan (TCDB I) with at least one risk factor :

  * GCS = 14 after CT scan
  * and/or alcoholic intoxication
  * and/or on-going treatment with anticoagulants or anti-platelet therapy
  * and /or persisting nausea, and/or vomiting and/or headaches
  * Early initial CT scan (< 4 hours after TBI)
* Possibility of home supervision by a third-party
* Affiliation to the French social security system
* Patient have signed consent form
* Possibility to perform a TCD within 12 hours
* Stable hemodynamics defined as a blood pressure greater than 90 mmHg, an SpO2 greater than 92% and a hemoglobin concentration greater than 8g/dl, or, in the absence of measured physiologic parameters or the absence of biological sampling, mention in the patient's medical record of a stable clinical examination in terms of hemodynamics and respiratory function.

Exclusion Criteria:

* CT scan classified as TCDB III - VI
* Penetrating head-trauma
* Patient under mechanical ventilation
* Patients treated with anticoagulants or anti-platelet therapy (except Aspirin)
* Hospitalization required by post-traumatic extra-cranial lesion, intoxication (except alcoholic), pre-existing condition (including congenital hemostasis disorders) or social factors at the discretion of the physician.
* Internal Carotid dissection
* Post-traumatic lesion in the posterior cerebral fossa
* Subject in exclusion period of another interventional study,
* Pregnant women, breastfeeding women
* Subject under administrative or judicial control, under protection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of a TCD-based strategy after a mild TBI to the standard management in terms of the overall neurological outcome | 3 months after TBI
  GOS-E will be dichotomized as complete recovery (GOS-E 8) vs. incomplete recovery (GOS-E 1 to 7). Evaluation is centralized and blinded.

SECONDARY OUTCOMES:
Effects of a TCD-based strategy after a mild TBI on the overall neurological outcome | 1 month after TBI
  GOS-E will be dichotomized as complete recovery (GOS-E 8) vs. incomplete recovery (GOS-E 1 to 7). Evaluation is centralized and blinded.
Effects of a TCD-based strategy after a mild TBI on the quality of life | 1 months after TBI
  Questionnaires QOLIBRI (Quality of life after TBI) and EQ-5D-5L
Effects of a TCD-based strategy after a mild TBI on the quality of life | 3 months after TBI
  Questionnaires QOLIBRI (Quality of life after TBI) and EQ-5D-5L
Effects of a TCD-based strategy after a mild TBI on Post-concussive syndrome | 1 month after TBI
  Rivermead Post-Concussion Symptoms questionnaire at 1 month and 3 months after TBI ("Rivermead positive" patients are patients with at least 3 symptoms rated ≥ 2)
Effects of a TCD-based strategy after a mild TBI on Post-concussive syndrome | 3 months after TBI
  Rivermead Post-Concussion Symptoms questionnaire at 1 month and 3 months after TBI ("Rivermead positive" patients are patients with at least 3 symptoms rated ≥ 2)
Effects of a TCD-based strategy after a mild TBI on mortality after TBI | 3 months after TBI
  Mortality within the first 3 months
Effects of a TCD-based strategy after a mild TBI on Morbidity after TBI | 1 months after TBI
  Number of cerebral CT scans within the hospital stay, • Thromboembolic events or diagnosed nosocomial infections stay
Effects of a TCD-based strategy after a mild TBI on Morbidity after TBI | 1 months after TBI
  Length of hospital stay ; Length of ICU stay
Effects of a TCD-based strategy after a mild TBI on patient safety | 1 months after TBI
  Number of patients re-admitted to hospital in relation with the initial TBI
Effects of a TCD-based strategy after a mild TBI on patient safety | 3 months after TBI
  Number of patients with neurologic worsening within the first week after TBI.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUZAT, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (12):
- France (12):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble Alpes, Grenoble
  - HCL - Edouard Herriot, Lyon
  - HCL - Lyon Sud, Lyon
  - CH Melun, Melun
  - CHU Nantes, Nantes
  - AP-HP Lariboisière, Paris
  - AP-HP Pitié Salpetrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Réunion, Saint-Denis
  - Chu Reunion, Saint-Pierre
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maas AIR, Menon DK, Adelson PD, Andelic N, Bell MJ, Belli A, Bragge P, Brazinova A, Buki A, Chesnut RM, Citerio G, Coburn M, Cooper DJ, Crowder AT, Czeiter E, Czosnyka M, Diaz-Arrastia R, Dreier JP, Duhaime AC, Ercole A, van Essen TA, Feigin VL, Gao G, Giacino J, Gonzalez-Lara LE, Gruen RL, Gupta D, Hartings JA, Hill S, Jiang JY, Ketharanathan N, Kompanje EJO, Lanyon L, Laureys S, Lecky F, Levin H, Lingsma HF, Maegele M, Majdan M, Manley G, Marsteller J, Mascia L, McFadyen C, Mondello S, Newcombe V, Palotie A, Parizel PM, Peul W, Piercy J, Polinder S, Puybasset L, Rasmussen TE, Rossaint R, Smielewski P, Soderberg J, Stanworth SJ, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Synnot A, Te Ao B, Tenovuo O, Theadom A, Tibboel D, Videtta W, Wang KKW, Williams WH, Wilson L, Yaffe K; InTBIR Participants and Investigators. Traumatic brain injury: integrated approaches to improve prevention, clinical care, and research. Lancet Neurol. 2017 Dec;16(12):987-1048. doi: 10.1016/S1474-4422(17)30371-X. Epub 2017 Nov 6. No abstract available. PMID 29122524
- [Background] Tagliaferri F, Compagnone C, Korsic M, Servadei F, Kraus J. A systematic review of brain injury epidemiology in Europe. Acta Neurochir (Wien). 2006 Mar;148(3):255-68; discussion 268. doi: 10.1007/s00701-005-0651-y. PMID 16311842
- [Background] Davis DP, Kene M, Vilke GM, Sise MJ, Kennedy F, Eastman AB, Velky T, Hoyt DB. Head-injured patients who "talk and die": the San Diego perspective. J Trauma. 2007 Feb;62(2):277-81. doi: 10.1097/TA.0b013e31802ef4a3. PMID 17297312
- [Background] af Geijerstam JL, Britton M. Mild head injury: reliability of early computed tomographic findings in triage for admission. Emerg Med J. 2005 Feb;22(2):103-7. doi: 10.1136/emj.2004.015396. PMID 15662058
- [Derived] Bouzat P, Gauss T, Adolle A, Roustit M, Bosson JL, Tazarourte K. Transcranial Doppler to guide early discharge after mild traumatic brain injury, the TRUST trial: study protocol for an open-label multisite noninferiority randomized controlled trial. Trials. 2025 Sep 29;26(1):371. doi: 10.1186/s13063-025-09086-0. PMID 41024218